CLINICAL TRIAL: NCT05241639
Title: Pentacam Study of Rheumatoid Arthritis Activity on Corneal Densitometry, Corneal Curvature, Corneal Thickness and Lens Densitometry.
Brief Title: Pentacam Study of the Cornea in RA Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Dr Mohamed Salah, Minia University
Other Study IDs: 632-6/2020.
Record Dates: First submitted 2022-02-04; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: RA - Rheumatoid Arthritis
Keywords: Pentacam-RA-Corneal densitometry
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: of RA in the remission state
  Interventions: Diagnostic Test: Pentacam
- group 2: of RA in the active state
  Interventions: Diagnostic Test: Pentacam
- Group 3: 120 eyes of healthy controls.
  Interventions: Diagnostic Test: Pentacam

INTERVENTIONS:
Diagnostic Test: Pentacam — Pentacam (Oculus GmbH, Wetzlar, Germany) is used to image both the anterior and posterior corneal surfaces, providing a complete pachymetry map. Furthermore, it includes the corneal densitometry program in its software, which detects the amount of backscattered light in different regions of the cornea, providing an objective assessment of corneal transparency, and it is hypothesized that corneal densitometry may be altered in the presence of a systemic inflammatory disease, even in the absence of any corneal haze or scar

SUMMARY:
To evaluate the effect of rheumatoid arthritis (RA) activity on the corneal densitometry, corneal curvature (CC), central corneal thickness (CCT), and lens densitometry by Pentacam and compared these parameters with those of age-matched healthy control subjects

DETAILED DESCRIPTION:
Case - control observational study on RA patients which divided into 2 groups, each group 120 eyes of 60 patients, group 1 of RA in the remission state and group 2 of RA in the active state. Group 3 of 120 eyes of healthy controls. Pentacam was used to measure corneal densitometry, CC, CCT, and lens densitometry. The cornea was divided into 4 concentric zones (0-2, 2-6, 6-10, and 10-12) and anterior, central, and posterior layers according to the depth

ELIGIBILITY:
Inclusion Criteria:

* The included patients had aged more than 20 years with RA only without ocular manifestations with clinically clear cornea with normal anterior and posterior segment examinations with normal intraocular pressure (IOP)

Exclusion Criteria:

* We excluded patients with ocular problems as corneal opacity, cataract, glaucoma, errors of refraction, topical application of eye drops except for topical artificial tears. The presence of systemic diseases other than RA as DM, hypertension were also excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study subjects were divided into 3 groups, group 1 of 120 eyes of 60 RA patients with disease remission, group 2 of 120 eyes of 60 RA patients with disease activity and group 3 of 120 eyes of 60 healthy group 3 of similar age group.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-05-13 (Estimated); Study Completion 2022-05-13 (Estimated)

PRIMARY OUTCOMES:
Corneal densitometry | through study completion, an average of 1 year".
  The central zone was a 2-mm-diameter circle located around the corneal apex. The second zone was shaped as an annulus situated 2-6 mm peripheral to the central zone. The annulus extending from 6-10 mm was the third zone. The fourth zone was the outermost zone and extended from 10-12 mm. The cornea is also subdivided based on depth into 3 different layers: anterior (the superficial 120 um), posterior (the innermost 60 um), and central (between these 2 layers).
Corneal thickness | through study completion, an average of 1 year".
  central corneal thickness
lens densitometry | through study completion, an average of 1 year".
  The mean densitometry value was calculated for the crystalline lens in three zones located around the pupil center comprising zone 1 (2.0 mm in diameter), zone 2 (4.0 mm in diameter), and zone 3 (6.0 mm in diameter).The lens densitometry was evaluated from scheimpflug images and the average lens opacity was used

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Mahmoud, Principal Investigator — Minia faculty of medicine
Locations (2):
- Egypt (2):
  - Minia Faculty of medicine, Minya
  - Minia University hospital, Minya

IPD SHARING:
Plan to Share IPD: No
IPD arenot to be shared with other researchers.